CLINICAL TRIAL: NCT04964804
Title: Comparative Study of Real-time Ultrasound-CT Fusion Imaging and Ultrasound-guided Selective Lumbar Nerve Root Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2016207
Record Dates: First submitted 2021-06-27; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real-time ultrasound-CT fusion imaging (Experimental): The experimental group of patients underwent selective lumbar nerve root block puncture under real-time ultrasound-CT fusion imaging by sonographers
  Interventions: Procedure: real-time ultrasound-CT fusion imaging
- ultrasound alone (Active Comparator): The control group underwent puncture under the guidance of ultrasound alone by sonographers
  Interventions: Procedure: ultrasound alone

INTERVENTIONS:
Procedure: real-time ultrasound-CT fusion imaging — selective lumbar nerve root block puncture under real-time ultrasound-CT fusion imaging
  Arms: real-time ultrasound-CT fusion imaging
Procedure: ultrasound alone — selective lumbar nerve root block puncture under the guidance of ultrasound alone
  Arms: ultrasound alone

SUMMARY:
The study is aimed at patients with low back and leg pain. The experimental group of patients underwent selective lumbar nerve root block puncture under real-time ultrasound-CT fusion imaging by sonographers, and the control group underwent puncture under the guidance of ultrasound alone by sonographers.

DETAILED DESCRIPTION:
A total of 60 patients with low back and leg pain were randomly divided into two groups, 30 people in each group. Patients in the experimental group underwent selective lumbar nerve root block puncture under the real-time ultrasound-CT fusion imaging of the sonographer, and the control group underwent puncture under the sole ultrasound guidance of the sonographer. This study was used to compare the difference between the effects of pure ultrasound guidance and ultrasound-CT fusion imaging guidance on selective lumbar nerve root block.

ELIGIBILITY:
Inclusion Criteria:

Patients who need lumbar nerve root block treatment

Exclusion Criteria:

1. Tumor patients
2. Patients who have had lumbar spine surgery before

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2016-05-14 (Actual)

PRIMARY OUTCOMES:
1 month VAS pain score | VAS pain scores were performed 1 month after surgery
  Patients undergo VAS pain score after the sonographer performs selective lumbar nerve root block puncture
3 month VAS pain score | VAS pain scores were performed 3 month after surgery
  Patients undergo VAS pain score after the sonographer performs selective
6 month VAS pain score | VAS pain scores were performed 6 month after surgery
  Patients undergo VAS pain score after the sonographer performs selective
12 month VAS pain score | VAS pain scores were performed 12 month after surgery
  Patients undergo VAS pain score after the sonographer performs selective

CONTACTS AND LOCATIONS:
Overall Officials: Jinrui Wang, Study Director — Peking University Third Hospital
Locations (1):
- Department of Ultrasound Diagnosis, Peking University Third Hospital, Beijing, Beijing Municipality, China